CLINICAL TRIAL: NCT06600360
Title: Accuracy of Teledentistry for Diagnosis and Treatment Need in Dental Caries Detection Versus Clinical Examination on a Group of Egyptian Children: A Diagnostic Accuracy Study
Status: Not yet recruiting | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Pancee Adel Abdel Aziz Wafi, Teaching Assistant at Faculty of Dentistry, NewGiza University
Other Study IDs: TELE24
Record Dates: First submitted 2024-09-13; First posted 2024-09-19 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Teledentistry
Keywords: Teledentistry in diagnosis and treatment planning; Teledentistry

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Teledentistry — Measuring the accuracy of the mobile photographic method of teledentistry for diagnosis and treatment need in dental caries detection

SUMMARY:
The aim of this study is to assess the accuracy of teledentistry for diagnosis and treatment need in dental caries detection versus clinical examination on a group of Egyptian children.

DETAILED DESCRIPTION:
The objective of this study is to assess the precision of using the mobile photographic method of teledentistry for dental caries diagnosis and treatment need of pediatric Egyptian children. This will be assessed by measuring the diagnostic accuracy of the mobile photographic method versus direct clinical oral examination for the same group of participants.

ELIGIBILITY:
Inclusion Criteria:

* Egyptian pediatric patients aged 4 to 12 years with a chief complaint of dental caries with or without pain.
* Both genders are included.

Exclusion Criteria:

* Egyptian pediatric patients with systemic conditions that will affect their treatment needs.
* Refusal of participation.
* Refusal to sign the informed consent.

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Participants are Egyptian children with dental caries attending the diagnostic center at the Pediatric Dentistry and Dental Public Health Department, Faculty of Dentistry, Cairo University, Egypt.
Sampling Method: Probability Sample
Enrollment: 102 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2025-09-15 (Estimated); Study Completion 2025-10-15 (Estimated)

PRIMARY OUTCOMES:
Teledentistry for dental caries detection | 3 months
  By measuring the accuracy of mobile photographic method of teledentistry for dental caries detection

SECONDARY OUTCOMES:
Clinical dental caries examination | 3 months
  By measuring the accuracy of clinical dental caries examination
Reliability of treatment needs | 3 months
  By measuring the accuracy of teledentistry for treatment need

IPD SHARING:
Plan to Share IPD: Undecided